CLINICAL TRIAL: NCT01585727
Title: Continuous Intraoperative Monitoring of the Pelvic Autonomic Nerves During Total Mesorectal Excision (TME) for the Prevention of Urogenital and Anorectal Dysfunction in Patients With Rectal Cancer.
Brief Title: Intraoperative Monitoring of the Pelvic Autonomic Nerves
Acronym: NEUROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Werner Kneist, Senior physician, Department of Visceral and Abdominal Surgery, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007-012; KN 930/1-1 (Other Grant/Funding Number: German Research Foundation (DFG))
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; total mesorectal excision; pelvic autonomic nerve preservation; neurostimulation; urogenital function; quality of life
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TME with neuromonitoring (Experimental): Total mesorectal excision with intraoperative neuromonitoring of pelvic autonomic nerves.
  Interventions: Procedure: TME; Procedure: Neuromonitoring
- TME without neuromontoring (Active Comparator): Total mesorectal excision without intraoperative neuromonitoring of pelvic autonomic nerves.
  Interventions: Procedure: TME

INTERVENTIONS:
Procedure: TME — Total mesorectal excision
  Arms: TME with neuromonitoring
Procedure: TME — Total mesorectal excision
  Arms: TME without neuromontoring
Procedure: Neuromonitoring — Intraoperative neuromonitoring of pelvic autonomic nerves.
  Arms: TME with neuromonitoring

SUMMARY:
One of the major problems of rectal cancer surgery is pelvic autonomic nerve damage, which is the main cause of urogenital dysfunction influencing postoperative quality of life. Costs for diagnostics and treatment of short and long-term urogenital dysfunction are immense. Varying degrees of urogenital dysfunction are found in up to 32% and 55% of patients with rectal cancer despite potentially nerve-sparing total mesorectal excision (TME).

The study will examine the impact of a newly developed continuous monitoring device for preservation of urogenital function in patients with TME for rectal cancer. 188 patients will be included in the prospective, randomized, single-blind, parallel group multi-centre trial including two arms (TME with and without intraoperative continuous monitoring of pelvic autonomic nerves). The primary efficacy endpoint is the change in urinary function measured by International Prostate Function Score (IPSS) 12 months after surgery. Genital functions measured as secondary endpoints. The application of the continuous intraoperative neuromonitoring device could enhance the objective intraoperative confirmation of pelvic nerve sparing surgery. The investigators hypothesis is that the use of his device minimizes the risk of postoperative urogenital dysfunction in patients with TME for rectal cancer. An enormous reduction of treatment costs is to be expected.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* histologically confirmed carcinoma of the rectum (≤ 16 cm from anal verge)
* fit for radical surgery
* total mesorectal excision
* age 18-80 years

Exclusion Criteria:

* history of operation of the urinary tract (e.g. prostatectomy)
* pacemaker
* emergency operation
* multivisceral resection in the pelvis
* partial mesorectal excision
* eligibility for local excision (TEM, intestinal wall resection)
* ongoing infection or sepsis
* severe untreated physical or mental impairment
* pregnancy or breastfeeding
* women of childbearing potential who are not using a highly effective birth control method
* missing preoperative data on urogenital or anorectal function
* simultaneous participation in another clinical trial
* previous participation in this clinical trial
* lack of cooperation with the trial procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-06; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Urogenital function | 12 months
  Increase of IPSS score by at least 5 points observed 12 months after surgery compared to the preoperative IPSS score per patient

SECONDARY OUTCOMES:
Sexual function (females) | 12 months
  Reduction of FSFI score by at least 8 points 12 months after surgery compared to the preoperative FSFI score per patient.
Sexual function (males) | 12 months
  Reduction of IIEF score by at least 15 points 12 months after surgery compared to the preoperative IIEF score per patient.
Adverse events | 12 months
  Occurrence of adverse events.
Oncological safety | 12 months
  Rates of pCRM-positive specimen (distance of tumour from circumferential resection margin (CRM) ≤ 1mm).
Quality of mesorectal excision | 1 day after the surgery
  Macroscopic assessment of the resection specimen.
Fecal incontinence | 12 months
  Evaluation of fecal incontinence using the Wexner-Vaizey score

CONTACTS AND LOCATIONS:
Overall Officials: Werner Kneist, Univ.-Prof., Principal Investigator — Department of Visceral and Abdominal Surgery, University Medical Center Mainz
Locations (1):
- Department of General and Visceral Surgery, University Medical Center Mainz, Mainz, Germany

REFERENCES:
- [Derived] Kauff DW, Kronfeld K, Gorbulev S, Wachtlin D, Lang H, Kneist W. Continuous intraoperative monitoring of pelvic autonomic nerves during TME to prevent urogenital and anorectal dysfunction in rectal cancer patients (NEUROS): a randomized controlled trial. BMC Cancer. 2016 May 21;16:323. doi: 10.1186/s12885-016-2348-4. PMID 27209237